CLINICAL TRIAL: NCT06428019
Title: A Prospective, Open-Label, Phase IIb/III Study to Evaluate the Risk of TLS and Optimization of the Initiation of Venetoclax in Combination With Obinutuzumab or Acalabrutinib With Different Ramp- Up Periods in Previously Untreated Subjects With CLL
Brief Title: A Study to Evaluate the Risk of Tumor Lysis Syndrome (TLS) in Adult Participants Receiving Oral Venetoclax in Combination With Intravenously Infused Obinutuzumab or Oral Acalabrutinib for Previously Untreated Chronic Lymphocytic Leukemia (CLL)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M24-287; 2024-512147-23-00 (Other: EU CT)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Venetoclax; ABT-199; Obinutuzumab; Acalabrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax; acalabrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm A: Venetoclax + Obinutuzumab (Experimental): Participants will receive venetoclax in combination with obinutuzumab, with a 5 week venetoclax ramp up.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab
- Arm B: Venetoclax + Acalabrutinib (Experimental): Participants will receive venetoclax in combination with acalabrutinib, with a 5 week venetoclax ramp up.
  Interventions: Drug: Venetoclax; Drug: Acalabrutinib
- Arm C: Venetoclax + Acalabrutinib (Experimental): Participants will receive venetoclax in combination with acalabrutinib, with a modified venetoclax ramp up A.
  Interventions: Drug: Venetoclax; Drug: Acalabrutinib
- Arm D: Venetoclax + Acalabrutinib (Experimental): Participants will receive venetoclax in combination with acalabrutinib, with a modified venetoclax ramp up B.
  Interventions: Drug: Venetoclax; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Venetoclax — Oral: Tablet
  Other Names: ABT-199
Drug: Acalabrutinib — Oral: Tablet
  Arms: Arm B: Venetoclax + Acalabrutinib; Arm C: Venetoclax + Acalabrutinib; Arm D: Venetoclax + Acalabrutinib
Drug: Obinutuzumab — Intravenous Infusion
  Arms: Arm A: Venetoclax + Obinutuzumab

SUMMARY:
Chronic lymphocytic leukemia (CLL) is the most common leukemia (cancer of blood cells). The purpose of this study is to assess the safety of venetoclax in combination with obinutuzumab or acalabrutinib in the treatment of CLL. Adverse events and change in disease activity will be assessed.

Venetoclax in combination with obinutuzumab or acalabrutinib is being investigated in the treatment of CLL. Study doctors put the participants in 1 of 4 groups, called treatment arms. Participants will receive oral venetoclax in combination with intravenously (IV) infused obinutuzumab or oral acalabrutinib at in different dosing schemes as part of treatment. Approximately 170 adult participants with CLL who are being treated with venetoclax will be enrolled in the study in approximately 80 sites worldwide.

Participants in Arm A will receive oral venetoclax in combination with IV infused obinutuzumab, with a 5 week venetoclax ramp up. Participants in Arm B will receive oral venetoclax in combination with oral acalabrutinib, with a 5 week venetoclax ramp up. Participants in Arm C and Arm D will receive oral venetoclax in combination with oral acalabrutinib, with differing venetoclax ramp up periods. The total study duration is approximately 28 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of documented, previously untreated, chronic lymphocytic leukemia (CLL) requiring treatment according to the 2018 international workshop on chronic lymphocytic leukemia (iwCLL) criteria and have a life expectancy of > 6 months.
* Previously untreated small lymphocytic lymphoma (SLL) meeting the 2018 iwCLL criteria for treatment will also be equally considered as CLL for eligibility, screening, treatment and evaluation.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2.
* Adequate marrow function independent of growth factor or transfusion support within 2 weeks of screening, unless cytopenia is due to marrow involvement of CLL as listed in the protocol.
* Creatinine clearance (CrCl) >= 30 mL/min using the Cockcroft-Gault formula are eligible for inclusion.

Exclusion Criteria:

- Active/uncontrolled infection, no Richter's transformation, no active immune thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Part 1: Percentage of Participants with Treatment-Emergent Laboratory Tumor Lysis Syndrome (TLS)-Venetoclax | Up to 28 Months
  TLS is defined per Howard criteria that require a clinical intervention per independent review committee (IRC) assessment during the venetoclax ramp-up period in previously untreated participants with chronic lymphocytic leukemia (CLL) achieving a medium tumor burden with creatinine clearance (CrCl) of at least 80 ml/min or low tumor burden (regardless of CrCl level) after debulking therapy.
Part 1: Percentage of Participants with Hyperkalemia-Venetoclax | Up to 28 Months
  Hyperkalemia (potassium >6.0 mmol/L) is defined per Howard criteria that require a clinical intervention per IRC assessment during the venetoclax ramp-up period in previously untreated participants with CLL achieving a medium tumor burden with CrCl of at least 80 ml/min or low tumor burden (regardless of CrCl level) after debulking therapy.

SECONDARY OUTCOMES:
Part 1: Percentage of Participants with Treatment-Emergent Laboratory TLS | Up to 28 Months
  TLS is defined per Howard criteria that require a clinical intervention per IRC assessment, at each dose level and at each laboratory monitoring point during ramp-up period in previously untreated participants with CLL achieving a medium tumor burden with CrCl of at least 80 ml/min or low tumor burden (regardless of CrCl level) after debulking therapy.
Part 1: Percentage of Participants with Hyperkalemia | Up to 28 Months
  Hyperkalemia (potassium >6.0 mmol/L) is defined per Howard criteria that require a clinical intervention per independent review committee (IRC) assessment during the venetoclax ramp-up period in previously untreated participants with CLL achieving a medium tumor burden with CrCl of at least 80 ml/min or low tumor burden (regardless of CrCl level) after debulking therapy.
Part 1: Percentage of Participants with Treatment-Emergent TLS-Related Events | Up to 28 Months
  TLS-related events are defined as laboratory TLS per Howard criteria requiring clinical intervention per IRC assessment, hyperkalemia (potassium >6.0 mmol/L) requiring clinical intervention per IRC assessment, laboratory TLS per Howard criteria irrespective of clinical intervention, Hyperkalemia (potassium >6.0 mmol/L) irrespective of clinical intervention, clinical TLS per Howard criteria irrespective of clinical intervention, any single TLS-related lab abnormality requiring clinical intervention per Investigator.
Part 1: Percentage of Participants with Adverse Events (AE) of TLS | Up to 28 Months
  AEs of TLS is defined as a blood chemistry changes or symptom suggestive of TLS.
Part 1: Percentage of Participants with Reduction of Tumor Burden from Baseline | Up to 28 Months
  Percentage of participants with reduction of tumor burden.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (70):
- United States (32):
  - Arizona Oncology - Tucson - Rudasill /ID# 267552, Tucson, Arizona
  - Southern VA Health Care System /ID# 266254, Tucson, Arizona
  - UCSF FRESNO/Community Cancer Institute /ID# 270874, Clovis, California
  - Valkyrie Clinical Trials /ID# 268151, Los Angeles, California
  - Rocky Mountain Cancer Centers - Aurora /ID# 267549, Aurora, Colorado
  - Yale University School of Medicine /ID# 266224, New Haven, Connecticut
  - Malcolm Randall V.A. Medical Center /ID# 267825, Gainesville, Florida
  - Cancer Specialists of North Florida - Jacksonville - AC Skinner Parkway /ID# 266713, Jacksonville, Florida
  - Mid Florida Hematology And Oncology Center /ID# 269159, Orange City, Florida
  - Comprehensive Hematology Oncology /ID# 267644, St. Petersburg, Florida
  - Springfield Clinic - First /ID# 270145, Springfield, Illinois
  - Northwest Cancer Center - Dyer Clinic /ID# 268478, Dyer, Indiana
  - University of Iowa Health Care /ID# 267206, Des Moines, Iowa
  - Willis-Knighton Medical Center /ID# 270569, Shreveport, Louisiana
  - Center for Cancer and Blood Disorders-American Oncology Partners of Maryland /ID# 266445, Bethesda, Maryland
  - Maryland Oncology Hematology - Silver Spring /ID# 267557, Silver Spring, Maryland
  - UMass Memorial Medical Center /ID# 270023, Worcester, Massachusetts
  - Henry Ford Hospital /ID# 270973, Detroit, Michigan
  - Saint Lukes Hospital of Kansas City /ID# 267270, Kansas City, Missouri
  - Icahn School of Medicine at Mount Sinai /ID# 266328, New York, New York
  - Atrium Health /ID# 267219, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 273142, Winston-Salem, North Carolina
  - Cleveland Clinic Main Campus /ID# 271292, Cleveland, Ohio
  - Oklahoma Cancer Specialists and Research Institute /ID# 267643, Tulsa, Oklahoma
  - Willamette Valley Cancer Institute and Research Center /ID# 266326, Eugene, Oregon
  - Lifespan Cancer Institute - Providence /ID# 266550, Providence, Rhode Island
  - Texas Oncology - Austin Midtown /ID# 268152, Austin, Texas
  - University of Texas - Southwestern Medical Center /ID# 266528, Dallas, Texas
  - Virginia Cancer Specialists - Gainesville /ID# 268155, Gainesville, Virginia
  - Vista Oncology - East Olympia /ID# 267337, Olympia, Washington
  - Northwest Medical Specialties Tacoma /ID# 266327, Tacoma, Washington
  - West Virginia University School of Medicine /ID# 267645, Morgantown, West Virginia
- Australia (4):
  - Calvary Mater Newcastle /ID# 267408, Waratah, New South Wales
  - Townsville University Hospital /ID# 266954, Townsville, Queensland
  - St Vincent's Hospital - Melbourne /ID# 270027, Fitzroy, Victoria
  - Royal Perth Hospital /ID# 266906, Perth, Western Australia
- France (10):
  - Centre Hospitalier Régional Metz Thionville - Hôpital de Mercy /ID# 266852, Metz, Moselle
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 266270, Créteil, Paris
  - Hopitaux Universitaires Paris Centre-Hopital Cochin /ID# 267438, Paris, Paris
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 266319, St-Priest-en-Jarez, Pays de la Loire Region
  - Centre Antoine-Lacassagne /ID# 266894, Nice, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de la Côte Basque /ID# 266847, Bayonne, Pyrenees-Atlantiques
  - Centre Hospitalier Métropole Savoie - Site Hôpital de Chambéry /ID# 266854, Chambéry, Savoie
  - CHU Amiens-Picardie Site Sud /ID# 266849, Amiens, Somme
  - Centre Hospitalier Régional d'Orléans - Hôpital de la Source /ID# 266272, Orléans
  - Centre Hospitalier d Argenteuil Victor Dupouy /ID# 266322, Argenteuil, Île-de-France Region
- Greece (5):
  - Olympion General Clinic /ID# 266819, Pátrai, Achaia
  - Evangelismos Hospital /ID# 266815, Athens, Attica
  - General Hospital of Athens Laiko /ID# 266813, Athens, Attica
  - University General Hospital Attikon /ID# 266814, Athens, Attica
  - University General Hospital of Alexandroupoli /ID# 266816, Alexandroupoli, Evros
- Pan American Center for Oncology Trials /ID# 266243, Rio Piedras, Puerto Rico
- Serbia (7):
  - Clinical Hospital Center Zvezdara /ID# 266560, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 266579, Belgrade, Beograd
  - Clinical Hospital Center - Bežanijska Kosa /ID# 266567, Belgrade, Beograd
  - University Clinical Center Nis /ID# 266580, Niš, Nisavski Okrug
  - University Clinical Center Kragujevac /ID# 266568, Kragujevac, Sumadijski Okrug
  - Institute for Oncology of Vojvodina /ID# 266556, Kamenitz, Vojvodina
  - University Clinical Center Vojvodina /ID# 266674, Novi Sad
- Spain (6):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 267164, Santiago de Compostela, A Coruna
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 266967, Majadahonda, Madrid
  - Clinica Universidad de Navarra - Pamplona /ID# 267762, Pamplona, Navarre
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 266969, Madrid
  - Hospital MD Anderson Cancer Center Madrid /ID# 267167, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 266968, Seville
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 267046, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 267017, Taipei City, Taipei
  - China Medical University Hospital /ID# 267018, Taichung
  - Linkou Chang Gung Memorial Hospital /ID# 267045, Taoyuan
- Nottingham City Hospital /ID# 266991, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-287